CLINICAL TRIAL: NCT04651621
Title: SMA Targeted Magnetic Stimulation Against Auditory Verbal Hallucinations
Acronym: SMA-AVH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SMA-AVH
Record Dates: First submitted 2020-11-06; First posted 2020-12-03 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Auditory Hallucination
MeSH Terms: conditions — Hallucinations

STUDY DESIGN:
Intervention Model Description: First phase is a cross-over with two randomized blinded sessions with either verum cTBS or sham with wash-out, for each participant, and a second open feasibility treatment phase with 5 sessions/day over four days for participants with distressing auditory verbal hallucinations
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical sham coil, masked by an independent person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Open label active cTBS (Experimental): Four consecutive days with 40s cTBS, 100% MT over the SMA, five times a day with 50 minutes between stimulations
  Interventions: Device: continuous theta burst stimulation over the SMA
- active cTBS (Experimental): One test session with 40s active cTBS, 100% MT, over the SMA in the initial double blind cross-over phase
  Interventions: Device: continuous theta burst stimulation over the SMA
- Sham cTBS (Sham Comparator): One test session with 40s sham cTBS, 100% MT, over the SMA in the initial double blind cross-over phase with a special sham coil that diverts the magnetic field to be only superficial
  Interventions: Device: sham continuous theta burst stimulation over the SMA

INTERVENTIONS:
Device: continuous theta burst stimulation over the SMA — Each cTBS session consists of bursts of three pulses delivered with a rate of 50 Hz, with bursts repeated at a rate of 5 Hz for a total duration of 40 seconds, summing up to 600 pulses, 100% of motor threshold (MT) and applied over bilateral SMA. The target is located in the anterior-posterior direction over the transition between pre-SMA and SMA proper, (cortical point where a vertical line will pass through the anterior commissure). The center of a figure-of-eight coil will be placed over the target, guided with neuronavigation equipment that utilizes the anatomical brain image from the pre-cTBS scanning session.
  Arms: Open label active cTBS; active cTBS
Device: sham continuous theta burst stimulation over the SMA — The same stimulation parameters but a concealed sham coil will be used with only superficial magnetic stimulation to mimic the sensation of the active stimulation
  Arms: Sham cTBS

SUMMARY:
Auditory verbal hallucinations (AVH) are prevalent among patients with psychiatric disorders. Not only being highly stressful and functionally impairing, AVH often persist despite treatment. Recent attempts to treat AVH with add-on repetitive transcranial magnetic stimulation (rTMS) when targeting the temporoparietal junction (TPJ), a language node in the brain, has gained limited success. The aim of this investigation is to reduce AVH with rTMS using continous theta-burst stimulation over a novel target, the supplementary motor area (SMA), in participants with frequent AVH, while also assessing potential neurophysiological mechanisms underlying the symptom.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the AVH group:

* Reported AVH with a minimum frequency of at least daily occurrence, with onset more than one month ago
* Stable psychopharmacological treatment past month

Inclusion criteria for the non-AVH control group

* Reporting no occurrences of AVH for the past year
* Stable psychopharmacological treatment past month

Inclusion criteria for the healthy control group

* No life-time occurrence of AVH
* No history of psychiatric disorders as assessed with a Mini-International Neuropsychiatric Interview (M.I.N.I.)

Exclusion Criteria:

* Ferromagnetic or electromagnetic implants that may pose a risk during magnetic resonance imaging (MRI) and/or cTBS
* A history of epilepsy
* Pregnancy
* Current substance use disorder or a history of alcohol use disorder as assessed with Alcohol Use Disorders Identification Test (AUDIT), Drug Use Disorders Identification Test (DUDIT), urine samples with test for illicit drugs and Phosphatidylethanol (PEth)
* Daily benzodiazepine use
* Factors that make the participant unlikely to be able to complete the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Amplitude on EEG in speech-listen task | 5-30 minutes after intervention
  Neurophysiological outcome of the blinded cross-over phase
Change on The Psychotic Symptom Rating Scales (PSYRATS) | 1 day after completion of open treatment phase
  Auditory Verbal Hallucination symptom interview, total score

SECONDARY OUTCOMES:
Finger tapping test | 5-30 minutes after intervention
  Computerized version of the finger tapping test from The Halstead-Reitan Neuropsychological Test Battery, performance
Double step saccade-task | 20-60 minutes after intervention
  Performance (Zimmermann et al Sci Rep, 2018).
Resting state functional magnetic resonance imaging (rsfMRI) | 1 day after completion of open treatment phase
  Resting state SMA connectivity change as measured with fMRI
Magnetic resonance spectroscopy (MRS) over the SMA quantifying glutamate and gamma-aminobutyric acid (GABA) and other metabolites | 1 day after completion of open treatment phase
  Prefrontal GABA and Glutamate concentration change as measured with a MEGA-PRESS magnetic resonance spectroscopy sequence following intervention.
Brief Psychiatric Rating Scale (BPRS) | 1 day after completion of open treatment phase
  Total score
App recorded ratings of auditory verbal hallucinations (AVH) | From first day of open treatment phase, and through one week after completion of treatment
  5 times a day randomized time points for app ratings of AVH

CONTACTS AND LOCATIONS:
Overall Officials: Robert Boden, MD, Principal Investigator — Uppsala University
Locations (1):
- Department of neuroscience, psychiatry, unit for Brain Stimulation and psychiatric clinical trials, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No